CLINICAL TRIAL: NCT04213521
Title: Visual Dependence and Multisensory Balance Exercise for Elderly
Brief Title: Visual Dependence and Multisensory Balance Exercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N20180725
Record Dates: First submitted 2019-12-19; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2018-07

CONDITIONS: Visual Dependence; Multisensory; Exercise; Training; Balance; Elderly
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multisensory balance training group (Experimental): The participants in the multisensory balance training group were provided with multiple-sensory balance exercises using visual, proprioceptive, and vestibular manipulations. The exercises involved movements of the eye, head, and body to stimulate the vestibular system-postural control exercises in different positions (feet together, tandem stance, and one leg stance), use of a soft surface to reduce the proprioceptive inputs, and exercises with closed eyes to deprive them of visual cues.
  Interventions: Other: Multisensory balance exercise; Other: Conventional balance exercise
- Conventional balance training group (Active Comparator): The participants in the Conventional balance training group performed conventional balance exercises, such as static and dynamic standing balance without altered sensory inputs.
  Interventions: Other: Conventional balance exercise

INTERVENTIONS:
Other: Multisensory balance exercise — Multisensory balance training describes a balance exercise incorporating individual sensory manipulation of vision, vestibular, proprioception and sensory integration.
  Arms: Multisensory balance training group
Other: Conventional balance exercise — such as static and dynamic standing balance without altered sensory inputs.

SUMMARY:
The study aimed to investigate the effectiveness of multisensory balance training on the levels of visual dependence and sensory organization capacity in community-dwelling older adults. Participants in the experimental group received multisensory balance training while those in the control group received conventional balance training without sensory manipulation.

DETAILED DESCRIPTION:
Older people often find it difficult to maintain balance with their eyes closed, which emphasizes the importance of vision. The greater influence of vision on orientation and balance has been observed by manipulating static and dynamic visual cues-for instance, tilting the frame of reference or moving visual scenes. Older people-particularly those prone to falls-have been reported to make significantly greater errors in subjective visual verticality and exhibit greater sway and continued center of gravity oscillation during and following visual disturbances. They also adopted hip strategies to restore balance in response to visual perturbation, indicating that they were unstable in the event of visual disturbance. These results indicate that older people may have higher levels of visual dependence than younger adults.

The underlying mechanism of visual dependence remains unclear. Visual dependence is considered a form of sensory reweighting deficit. In a situation of sensory conflict, the central nervous system must first recognize the discrepancy and reduce the weighting (suppress) of the inaccurate input while increasing the weighting of the input from the sensory systems that are deemed to provide more reliable information. This complex process of sensory organization is termed multiple-sensory reweighting and is vital in maintaining balance and orientation in a continuously changing and complex environment.

Studies have suggested that visual dependence could benefit from promoting desensitization and increased visual motion tolerance through visual adaptation and habituation exercises in vestibular rehabilitation. This may be because the majority of visually dependent adults have the comorbid symptom of visual vertigo. However, according to the National Audit Survey in the United States, one-third of patients with vestibular disorders and visual dependence lack signs and symptoms of dizziness or vertigo. Recent evidence has demonstrated that healthy older adults with greater levels of visual dependence did not have dizziness; therefore, it is unclear whether visual adaptation exercises can effectively reduce the degree of visual dependence in such people. However, visual dependence can be considered as a sensory reweighting deficit; therefore, multisensory balance training with manipulation of the visual, vestibular, and proprioceptive inputs could be an alternative for decreasing visual dependence through improving the integration and reweighting of sensory systems. In fact, multiple studies have documented that multisensory balance training improves mobility and balance in older adults with instability or a history of falls; however, few have investigated its effectiveness on visual dependence and in healthy elderly people. Therefore, the aim of the study was to investigate the effectiveness of multisensory balance training on the levels of visual dependence and sensory organization capacity in older adults.

ELIGIBILITY:
Inclusion Criteria:

* 1) age more than 60 years
* 2) able to walk continuously for 10 meters independently without aid
* 3) normal cognitive function with a Mini-Mental State Examination score more than 24
* 4) able to follow oral commands.

Exclusion Criteria:

* any medical condition or recent injury that could affect the assessment of balance.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Rod and Disc Test | Change from baseline to post-intervention at 4-8 weeks
  It is a computerized test which measures levels of visual dependence. Greater errors from true vertical indicates the greater levels of visual dependence.
Modified clinical test of sensory interaction in balance | Change from baseline to post-intervention at 4-8 weeks
  It assess the contribution of the visual, somatosensory, and vestibular systems to postural control.

SECONDARY OUTCOMES:
Chair sit and reach test | Change from baseline to post-intervention at 4-8 weeks
  It measures lower limb flexibility.
Five times sit to stand test | Change from baseline to post-intervention at 4-8 weeks
  It measures lower limb strength.
Berg balance scale | Change from baseline to post-intervention at 4-8 weeks
  It is used to objectively determine a patient's ability to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function. A total score of 56 indicates functional balance and but less than 45 indicates individuals may be at greater risk of falling.
The Activities specific Balance Confidence Scale | Change from baseline to post-intervention at 4-8 weeks
  It measures balance confidence level and contains 16 items scored on a range from 0% to 100%. The score of 0 indicates no confidence and 100 indicates full confidence.
Timed up and go test | Change from baseline to post-intervention at 4-8 weeks
  It measures functional mobility. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down. Normal healthy elderly usually complete the task in 10 seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more. A score of more than or equal to 14 seconds has been shown to indicate high risk of falls.
10 meters walk test | Change from baseline to post-intervention at 4-8 weeks
  It is a performance measure used to assess walking speed and walking capacity in meters per second over a short distance.

OTHER OUTCOMES:
mini mental state examination | During screening
  It is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive function. Any score of 24 or more (out of 30) indicates a normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points) or mild (19-23 points) cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Chun Lee, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
would like to share if other researchers officially request
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: applicants need to provide their research background, purposes and the reasons why they request IPD, principal investigator will review the applicants, affiliations and all the documents mentioned above.